CLINICAL TRIAL: NCT01611792
Title: Effects and Mechanisms of Specific Trunk Exercises in Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Sharon M. Henry, Professor, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIH/NCMRR/R01-HD040909
Record Dates: First submitted 2012-06-01; First posted 2012-06-05 (Estimated); Results first posted 2017-08-21 (Actual); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Low Back Pain
Keywords: Stabilization exercise; Strength and conditioning exercise; Physical therapy; Rehabilitation
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stabilization (Experimental)
  Interventions: Other: Stabilization exercise protocol
- Strengthening and Conditioning (Active Comparator)
  Interventions: Other: Strength and conditioning exercise protocol

INTERVENTIONS:
Other: Stabilization exercise protocol — The stabilization exercise protocol consists of exercises focused on improving the ability of trunk muscles to stabilize the spine, beginning with training to isolate the deeper abdominal muscles as well as deep dorsal trunk muscles. Then patients were progressed to exercises that added leverage of the limbs while maintaining the co-contraction of the deeper abdominal muscles and deep dorsal trunk muscles while breathing normally. Various positions (e.g., supine and quadruped positions) were used to challenge the patients based on their tolerance. Finally, patients were progressed to exercises in more functional positions that included tasks/activities that were reported as challenging and/or painful; patients performed the tasks at the speed demanded by the particular task. Maintenance of the co-contraction of deep trunk muscles was emphasized during these functional activities.
  Other Names: Trunk stabilization exercises; Segmental stabilization exercises
  Arms: Stabilization
Other: Strength and conditioning exercise protocol — This protocol contained trunk strengthening and endurance exercises. It consisted of 3 phases: 1) initial strengthening of trunk flexors/extensors in single plane movements, 2) trunk and lower-extremity stretching as well as progression of trunk-strengthening exercises to include multi-planar trunk movements. Aerobic exercises were progressed as tolerated and patient education about body biomechanics were reinforced, and 3) trunk-strengthening exercises under dynamic conditions (e.g., unstable support surface and in multi-planar trunk movements). During the 10 week protocol, exercises became more challenging, and each subject had to complete at least the first phase before moving onto the next phase in order to be included in post-testing analyses. There was no specific focus on the deep abdominal or deep dorsal trunk muscles during any of these exercises.
  Other Names: General trunk exercise; General strength training
  Arms: Strengthening and Conditioning

SUMMARY:
Low back pain affects 80% of Americans at some time during their lives. Although recovery usually occurs within 6 months, there is a 50% recurrence within one year's time. It has long been thought that poor control of trunk muscle may lead to abnormal forces across the spine, which then damage local spinal structures, thus, leading to low back pain. However, the investigators know little about the function of specific trunk muscles in healthy subjects during various activities of daily life. Furthermore, the precise muscle dysfunction associated with low back pain has not been well characterized at all. In addition, the investigators know little about which exercise protocol is most beneficial for particular subgroups of people with low back pain. Thus, the purposes of this study are to learn more about: 1) how trunk muscles are affected by low back pain; 2) which exercises might be most beneficial for people with certain kinds of low back pain; and 3) how these exercises influence trunk muscle function. By having a better understanding of which trunk muscles are affected by low back pain, rehabilitation specialists can design exercise programs and therapeutic interventions that are more specific and more effective.

ELIGIBILITY:
Inclusion Criteria:

* a history of chronic LBP with or without recurrences for a minimum of 12 months
* between 21 - 55 years of age
* able to stand and walk without assistance
* have an Oswestry Disability Score of 19% or higher

Exclusion Criteria:

* any major structural spinal deformity including scoliosis, kyphosis, or stenosis
* spinal fracture or dislocation
* osteoporosis
* ankylosing spondylitis
* rheumatoid arthritis
* disc herniation with corroborating clinical signs and symptoms
* serious spinal complications such as tumor or infection
* previous spinal surgery
* frank neurological loss, i.e., weakness and sensory loss
* pain or paresthesia below the knee
* etiology of LBP other than the lumbar spine, e.g., hip joint
* history of neurological disease which required hospitalization
* active treatment for cancer
* history of unresolved cancer
* pregnancy or less than 6 months post-partum or less than 6 months post weaning
* magnified symptom-behavior
* worker's compensation or disability case
* in litigation for the LBP problem
* have a BMI ≥ 30

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2003-03; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon M Henry, PT, PhD, Principal Investigator — University of Vermont
Locations (1):
- Human Motion Analysis Laboratory, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jones SL, Henry SM, Raasch CC, Hitt JR, Bunn JY. Individuals with non-specific low back pain use a trunk stiffening strategy to maintain upright posture. J Electromyogr Kinesiol. 2012 Feb;22(1):13-20. doi: 10.1016/j.jelekin.2011.10.006. Epub 2011 Nov 18. PMID 22100719
- [Background] Jacobs JV, Henry SM, Jones SL, Hitt JR, Bunn JY. A history of low back pain associates with altered electromyographic activation patterns in response to perturbations of standing balance. J Neurophysiol. 2011 Nov;106(5):2506-14. doi: 10.1152/jn.00296.2011. Epub 2011 Jul 27. PMID 21795622
- [Background] Stokes IA, Gardner-Morse MG, Henry SM. Abdominal muscle activation increases lumbar spinal stability: analysis of contributions of different muscle groups. Clin Biomech (Bristol). 2011 Oct;26(8):797-803. doi: 10.1016/j.clinbiomech.2011.04.006. Epub 2011 May 14. PMID 21571410
- [Background] Stokes IA, Gardner-Morse MG, Henry SM. Intra-abdominal pressure and abdominal wall muscular function: Spinal unloading mechanism. Clin Biomech (Bristol). 2010 Nov;25(9):859-66. doi: 10.1016/j.clinbiomech.2010.06.018. Epub 2010 Jul 23. PMID 20655636
- [Background] Jones SL, Henry SM, Raasch CC, Hitt JR, Bunn JY. Responses to multi-directional surface translations involve redistribution of proximal versus distal strategies to maintain upright posture. Exp Brain Res. 2008 May;187(3):407-17. doi: 10.1007/s00221-008-1312-1. Epub 2008 Feb 26. PMID 18299821
- [Background] Teyhen DS, Gill NW, Whittaker JL, Henry SM, Hides JA, Hodges P. Rehabilitative ultrasound imaging of the abdominal muscles. J Orthop Sports Phys Ther. 2007 Aug;37(8):450-66. doi: 10.2519/jospt.2007.2558. PMID 17877281
- [Background] Henry SM, Teyhen DS. Ultrasound imaging as a feedback tool in the rehabilitation of trunk muscle dysfunction for people with low back pain. J Orthop Sports Phys Ther. 2007 Oct;37(10):627-34. doi: 10.2519/jospt.2007.2555. PMID 17970410
- [Background] Anderson-Worth SG, Henry SM, Bunn JY. Use of real time ultrasound feedback enhances learning the abdominal hollowing exercise in patients with low back pain. New Zealand J Physiotherapy. 35(1):4-11, 2007.
- [Background] Henry SM, Hitt JR, Jones SL, Bunn JY. Decreased limits of stability in response to postural perturbations in subjects with low back pain. Clin Biomech (Bristol). 2006 Nov;21(9):881-92. doi: 10.1016/j.clinbiomech.2006.04.016. Epub 2006 Jun 27. PMID 16806618
- [Background] Henry SM, Westervelt KC. The use of real-time ultrasound feedback in teaching abdominal hollowing exercises to healthy subjects. J Orthop Sports Phys Ther. 2005 Jun;35(6):338-45. doi: 10.2519/jospt.2005.35.6.338. PMID 16001905
- [Background] Lomond KV, Henry SM, Hitt JR, DeSarno MJ, Bunn JY. Altered postural responses persist following physical therapy of general versus specific trunk exercises in people with low back pain. Man Ther. 2014 Oct;19(5):425-32. doi: 10.1016/j.math.2014.04.007. Epub 2014 Apr 24. PMID 24853255

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Back Pain: Stabilization
  Stabilization exercise protocol: The stabilization exercise protocol consists of exercises focused on improving the ability of trunk muscles to stabilize the spine, beginning with training to isolate the deeper abdominal muscles as well as deep dorsal trunk muscles. Then patients were progressed to exercises that added leverage of the limbs while maintaining the co-contraction of the deeper abdominal muscles and deep dorsal trunk muscles while breathing normally. Various positions (e.g., supine and quadruped positions) were used to challenge the patients based on their tolerance. Finally, patients were progressed to exercises in more functional positions that included tasks/activities that were reported as challenging and/or painful; patients performed the tasks at the speed demanded by the particular task. Maintenance of the co-contraction of deep trunk muscles was emphasized during these functional activities.
Period: Initial Period: Time 0
Arm/Group | Low Back Pain | Strengthening and Conditioning
Started | 29 | 29
Completed | 17 | 20
Not Completed | 12 | 9
Not completed — unable to schedule 10 consecutive appts | 12 | 9
Period: Follow-up: at 11 Weeks
Arm/Group | Low Back Pain | Strengthening and Conditioning
Started | 17 | 20
Completed | 17 | 20
Not Completed | 0 | 0
Period: Followup: at 6 Months
Arm/Group | Low Back Pain | Strengthening and Conditioning
Started | 17 | 20
Completed | 11 | 7
Not Completed | 6 | 13
Not completed — Lost to Follow-up | 6 | 13

BASELINE CHARACTERISTICS:
Population: Based on subjects who completed the 10 week treatment protocol
Groups:
- Stabilization: Stabilization
  Stabilization exercise protocol: The stabilization exercise protocol consists of exercises focused on improving the ability of trunk muscles to stabilize the spine, beginning with training to isolate the deeper abdominal muscles as well as deep dorsal trunk muscles. Then patients were progressed to exercises that added leverage of the limbs while maintaining the co-contraction of the deeper abdominal muscles and deep dorsal trunk muscles while breathing normally. Various positions (e.g., supine and quadruped positions) were used to challenge the patients based on their tolerance. Finally, patients were progressed to exercises in more functional positions that included tasks/activities that were reported as challenging and/or painful; patients performed the tasks at the speed demanded by the particular task. Maintenance of the co-contraction of deep trunk muscles was emphasized during these functional activities.
- Total: Total of all reporting groups
Arm/Group | Stabilization | Strengthening and Conditioning | Total
Number analyzed (Participants) | 17 | 20 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 20 | 37
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (8.3) | 41.2 (7.9) | 40.9 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 8 | 9 | 17
Region of Enrollment [Number; unit: participants]
  United States | 17 | 20 | 37
Numeric Pain Index [Mean (Standard Deviation); unit: units on a scale] — Current Pain; Scale 0-10; Lower score is better/improved; Collected on paper; patient self-report
  units on a scale | 3.7 (1.7) | 3.2 (1.5) | 3.2 (1.3)
Modified Oswestry Disability Index [Mean (Standard Deviation); unit: units on a scale] — Disability; Sacle 0-100%; Lower score is considered better/improve; Collected on paper; patient self-report
  units on a scale | 22.3 (9.7) | 20.1 (7.8) | 20.8 (8.4)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 11 Weeks in Oswestry Disability Scale (0-100%)
Description: Disability; Scale 0-100% Lower score is considered better/improved Negative value indicates improvement
Time Frame: Baseline and 11 weeks
Population: Based on data reported and available
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stabilization | Strengthening and Conditioning
Number analyzed (Participants) | 17 | 20
units on a scale | -11.06 (7.45) | -9.10 (10.27)
Statistical Analysis 1: Comparison: Stabilization vs Strengthening and Conditioning; Test type: Superiority; p < .0001, Mixed Models Analysis; Mean Difference (Net) = -10.0, Standard Deviation 9.02

2. Primary Outcome: Change From Baseline to 6 Months in Oswestry Disability Scale (0-100%)
Description: Disability; Sacle 0-100% Lower score is considered better/improved; Negative value indicates improvement
Time Frame: Baseline and 6 Months
Population: Based on data reported and available
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stabilization | Strengthening and Conditioning
Number analyzed (Participants) | 11 | 7
units on a scale | -10.73 (9.73) | -0.29 (12.78)
Statistical Analysis 1: Comparison: Stabilization vs Strengthening and Conditioning; Test type: Superiority; p = 0.0038, Mixed Models Analysis; Mean Difference (Net) = -6.67, Standard Deviation 11.86

3. Primary Outcome: Change From 11 Weeks to 6 Months in Oswestry Disability Scale (0-100%)
Description: Disability; Sacle 0-100% Lower score is considered better/improved; Negative value indicates improvement
Time Frame: 11 Weeks and 6 Months
Population: Based on data reported and available
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stabilization | Strengthening and Conditioning
Number analyzed (Participants) | 11 | 7
units on a scale | 0.55 (4.12) | 4.29 (6.58)
Statistical Analysis 1: Comparison: Stabilization vs Strengthening and Conditioning; Test type: Superiority; p = 0.36, Mixed Models Analysis; Mean Difference (Net) = 2.0, Standard Deviation 5.36

4. Primary Outcome: Change From Baseline to 11 Weeks in Numeric Pain Rating Scale (0-10 Points)
Description: Current Pain Scale 0-10 Lower score is better/improved; Negative value indicates improvement
Time Frame: Baseline and 11 weeks
Population: Based on data reported and available
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stabilization | Strengthening and Conditioning
Number analyzed (Participants) | 12 | 17
units on a scale | -0.67 (2.19) | -1.76 (1.75)
Statistical Analysis 1: Comparison: Stabilization vs Strengthening and Conditioning; Test type: Superiority; p = 0.0018, Mixed Models Analysis; Mean Difference (Net) = -1.31, Standard Deviation 1.98

5. Primary Outcome: Change From Baseline to 6 Months in Numeric Pain Rating Scale (0-10 Points)
Description: Current Pain Scale 0-10 Lower score is better/improved; Negative value indicates improvement
Time Frame: Baseline and 6 months
Population: Based on data reported and available
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stabilization | Strengthening and Conditioning
Number analyzed (Participants) | 10 | 6
units on a scale | -0.2 (1.6) | 2.2 (2.14)
Statistical Analysis 1: Comparison: Stabilization vs Strengthening and Conditioning; Test type: Superiority; p = 0.19, Mixed Models Analysis; Mean Difference (Net) = 0.69, Standard Deviation 2.12

6. Primary Outcome: Change From 11 Weeks to 6 Months in Numeric Pain Rating Scale (0-10 Points)
Description: Current Pain Scale 0-10 Lower score is better/improved; Negative value indicates improvement
Time Frame: 11 weeks and 6 months
Population: Based on data reported and available
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stabilization | Strengthening and Conditioning
Number analyzed (Participants) | 10 | 6
units on a scale | -0.2 (1.6) | 2.2 (2.1)
Statistical Analysis 1: Comparison: Stabilization vs Strengthening and Conditioning; Test type: Superiority; p = 0.19, Mixed Models Analysis; Mean Difference (Net) = 0.69, Standard Deviation 2.12

ADVERSE EVENTS:
Time Frame: From Baseline to completion of study
Arm/Group | Stabilization | Strengthening and Conditioning
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 0/29 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No